CLINICAL TRIAL: NCT00927147
Title: Boronophenylalanine (BPA)-Based Boron Neutron Capture Therapy (BNCT) Combined With Anti-erbB1 Antibody Therapy in the Treatment of Locally Recurred Head and Neck Cancer: A Phase I/II Study.
Brief Title: Boron Neutron Capture Therapy (BNCT) Combined With Cetuximab in the Treatment of Locally Recurred Head and Neck Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The neutron facility closed down for financial reasons.
Sponsor: Boneca Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN-BPA-01-2008
Record Dates: First submitted 2009-06-21; First posted 2009-06-24 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; boron neutron capture therapy; cetuximab; epidermal growth factor receptor; safety; efficacy; survival
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BNCT plus cetuximab (Experimental): Patients treated with BNCT followed by cetuximab administration
  Interventions: Radiation: BNCT; Drug: cetuximab

INTERVENTIONS:
Radiation: BNCT — Boronophenylalanine infusion followed by neutron irradiation
Drug: cetuximab — cetuximab infusion 250 to 400 mg/kg intravenously, 1 to 3 infusions
  Other Names: Erbitux

SUMMARY:
The purpose of the study is to investigate efficacy and safety boron neutron capture therapy (BNCT) administered in combination with cetuximab in the treatment of head and neck cancer that has recurred locally following conventional cancer treatment (surgery and radiation therapy). Boron neutron capture therapy is a special form of radiation therapy, which is based on interaction between boron atoms taken up by the cancerous tissue and neutron irradiation. The boron atoms, located within cancer cells, may capture low-energy neutrons obtained from a nuclear accelerator, which results in splitting up (fission) of the boron atoms, and a high radiation effect within the tumor. Cetuximab is an antibody directed against certain proteins found on cancer cell surface (epidermal growth factor receptors). When administered immediately after BNCT, cetuximab may or may not improve treatment efficacy.

DETAILED DESCRIPTION:
This is a single-center, non-randomized, non-comparative, open-label, phase I/II trial to determine safety and efficacy of BNCT in the treatment of nonoperable, irradiated, locally advanced cancers of the head and neck region. Patients will be treated with a single-fraction boronophenylalanine (BPA)-based BNCT. All patients will be evaluated for response using CT or magnetic resonance imaging (MRI).

Neutron irradiation will first be planned based on the available tumor imaging examinations, following which the head and body position will be determined for irradiation, and head fixation will be prepared and tested. On the irradiation day 400 mg/m2 L-BPA-F will be infused intravenously over 2 hours. Cetuximab doses will be administered following completion of BNCT. The cetuximab doses will be escalated in cohorts of 3 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive squamous cell carcinoma of the head and neck
* Inoperable tumor or the patient is not a candidate for surgery for medical reasons; prior surgery may or may not have been done
* Prior radiotherapy or chemoradiotherapy has been given to the tumor
* If prior 18F-boronophenylalanine (BPA) PET (positron emission tomography)has been done, BPA needs to accumulate at least 2 times more in the tumor than in the corresponding normal tissue
* A written informed consent

Exclusion Criteria:

* Presence of distant metastases
* A non-experimental, effective treatment op-tion is available
* WHO performance status >3
* WBC <2,500/mm3, platelets <75,000/mm3, serum creatinine >180 umol/L
* Concomitant systemic cancer chemotherapy (except cetuximab).
* Other concurrent experimental therapy
* Less than 1 month since prior radiation therapy
* Untreated or severe treated congestive heart failure or renal failure
* A cardiac pace-maker or unremovable metal implants present in the head and neck region that will interfere with MRI-based dose-planning
* Restlessness or inability to lie in a cast for 30 to 60 minutes
* Clinical follow-up after therapy cannot be arranged or the patient is not willing to participate in follow-up
* Pregnancy
* Age less than 18
* Known allergy/hypersensitivity to cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Response rate | December 2010

SECONDARY OUTCOMES:
Safety | December 2010
Duration of treatment response | December 2010
Time to progression | December 2010
Survival | December 2010
Adverse events | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Joensuu, MD, Study Chair — Department of Oncology, Helsinki University Central Hospital
Locations (1):
- Department of Oncology, Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Background] Kankaanranta L, Seppala T, Koivunoro H, Saarilahti K, Atula T, Collan J, Salli E, Kortesniemi M, Uusi-Simola J, Makitie A, Seppanen M, Minn H, Kotiluoto P, Auterinen I, Savolainen S, Kouri M, Joensuu H. Boron neutron capture therapy in the treatment of locally recurred head and neck cancer. Int J Radiat Oncol Biol Phys. 2007 Oct 1;69(2):475-82. doi: 10.1016/j.ijrobp.2007.03.039. Epub 2007 Aug 6. PMID 17689034